CLINICAL TRIAL: NCT00006052
Title: A Study to Determine the Efficacy and Safety of STI571 in Patients With Chronic Myeloid Leukemia in Accelerated Phase
Brief Title: STI571 in Treating Patients With Accelerated Phase Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000068087; NOVARTIS-STI5710114; MSKCC-00094
Record Dates: First submitted 2000-07-05; First posted 2004-04-02 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Leukemia
Keywords: accelerated phase chronic myelogenous leukemia; chronic myelogenous leukemia, BCR-ABL1 positive; Philadelphia chromosome negative chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: imatinib mesylate

SUMMARY:
RATIONALE: STI571 may interfere with the growth of cancer cells and may be effective treatment for chronic myelogenous leukemia.

PURPOSE: Phase II trial to study the effectiveness of STI571 in treating patients who have accelerated phase chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety of STI571 in patients with accelerated phase Philadelphia chromosome positive (or chromosome negative and Bcr/Abl positive) chronic myelogenous leukemia. II. Determine the rate of hematological response to this treatment in these patients. III. Determine the improvements in symptomatic parameters with this treatment in these patients. IV. Determine the cytogenetic response to this treatment in these patients. V. Determine the time to treatment failure in these patients after receiving this treatment.

OUTLINE: Patients receive oral STI571 daily. Treatment continues for at least 1 year in the absence of disease progression or unacceptable toxicity. Patients who are considered to have benefited may continue treatment beyond 1 year.

PROJECTED ACCRUAL: Not determined

ELIGIBILITY:
DISEASE CHARACTERISTICS: Confirmed diagnosis of chronic myelogenous leukemia in accelerated phase At least 15% but less than 30% blasts in blood or bone marrow At least 30% blasts plus promyelocytes in the peripheral blood or bone marrow At least 20% peripheral basophils Thrombocyte count less than 100,000/mm3 (unrelated to therapy) Patients must have never been in blastic phase Ph chromosome positive OR Ph chromosome negative and Bcr/Abl positive

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-3 Life expectancy: Not specified Hematopoietic: See Disease Characteristics Blood counts recovered from any prior antileukemic agents Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) (no greater than 3 times ULN if liver involvement suspected) AST and ALT no greater than 3 times ULN (no greater than 5 times ULN if liver involvement suspected) Renal: Creatinine no greater than 2 times ULN Cardiovascular: No grade 3 or 4 cardiac disease Other: No serious other concurrent medical condition Not pregnant or nursing Negative pregnancy test Fertile patients must use effective barrier contraception during and for at least 2 weeks after study for women and at least 3 months after study for men No history of noncompliance with medical regimens

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 48 hours since prior interferon alfa Prior hematopoietic stem cell transplantation allowed if blood counts have recovered No concurrent biologic therapy Chemotherapy: At least 14 days since prior homoharringtonine At least 24 hours since prior hydroxyurea At least 7 days since prior low dose cytarabine (less than 30 mg/m2 every 12-24 hours daily) At least 14 days since prior moderate dose cytarabine (100-200 mg/m2 for 5-7 days) At least 28 days since prior high dose cytarabine (1-3 g/m2 every 12-24 hours for 6-12 doses) At least 21 days since prior anthracyclines, mitoxantrone, etoposide, methotrexate, or cyclophosphamide At least 6 weeks since prior busulfan No concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified Other: At least 28 days since prior other investigational agents No concurrent other investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-06; Primary Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Monteleone, Study Chair — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals Corporation, East Hanover, New Jersey, United States